CLINICAL TRIAL: NCT06961669
Title: An Early Exploratory Clinical Study of Enhanced Autologous CAR-T Cell Injection (ECAR01) Targeting CD19 and BCMA in Patients With Relapsed or Refractory Multiple Myeloma, Acute B-Cell Leukemia, and B-Cell Lymphoma
Brief Title: Intravenous Autologous CD19 CAR-T Cells for R/ R MM, B-ALL, and B-Cell Lymphoma
Acronym: ECAR01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SWKCAR-T2024062401
Record Dates: First submitted 2025-04-22; First posted 2025-05-08 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Lymphoblastic Leukemia; Relapsed or Refractory Multiple Myeloma (RRMM)
Keywords: B-cell lymphoma; Relapsed or Refractory Multiple Myeloma; Acute B-Cell Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Multiple Myeloma; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Anti-BCMA and CD19 CART (Experimental): Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CART infusion. A dose of Anti-BCMA and CD19 CART will be infused on day 0.
  Interventions: Drug: Anti-BCMA and CD19 CART cells will be injected intravenously on a one-time basis

INTERVENTIONS:
Drug: Anti-BCMA and CD19 CART cells will be injected intravenously on a one-time basis — A single intravenous infusion of anti-BCMA and CD19 CART cells (dose-escalating infusion of 1.0-5.0 x10^5 CART cells/kg）.

SUMMARY:
This is an open label, single-site, dose-escalation study in up to 18 participants with Relapsed or Refractory Multiple Myeloma, Acute B-Cell Leukemia, and B-Cell Lymphoma. This study aims to evaluate the safety and efficacy of the treatment with Anti-BCMA and CD19 CART

ELIGIBILITY:
Inclusion Criteria:

1. The patient or his/her guardian is fully informed and agrees to participate in this clinical study and signs the informed consent form;
2. At the time of signing the informed consent form, be over 3 years of age, regardless of gender;
3. Patients with a confirmed diagnosis of acute B-cell leukemia/B-cell lymphoma/multiple myeloma who meet one of the following criteria:

   1. B diffuse large B-cell lymphoma (DLBCL), germinal center, or activated B-cell type; Primary cutaneous DLBCL; Primary mediastinal (thymic) large B-cell lymphoma; ALK anaplastic large B-cell lymphoma; High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement (i.e., "double or triple hit"); High-grade B-cell lymphoma; T-cell-rich B-cell lymphoma; transformed follicular lymphoma; or any aggressive B-cell lymphoma caused by indolent lymphoma; follicular lymphoma; mantle cell lymphoma; Patients with large cell transformation (Richter's Transformation) with CLL who have not achieved remission or have progressed after achieving remission after at least 1 prior line of therapy.
   2. Patients diagnosed with acute B-cell leukemia: Patients who have achieved relapse after achieving remission after prior chemotherapy; or patients who have failed to achieve remission (<5% bone marrow blasts or persistent extramedullary or central nervous system disease) after 2 prior cycles of induction chemotherapy, or who still maintain MRD.
   3. Multiple Myeloma: Patients with confirmed diagnosis of multiple myeloma and patients with relapsed or refractory multiple myeloma according to IMWG 2016 diagnostic criteria.
4. For patients with B-cell lymphoma, according to the recommendations for initial evaluation, staging, and response evaluation of Hodgkin and non-Hodgkin lymphoma (2014 edition), at least one measurable lesion in the baseline period, i.e., lymph node lesions with a length diameter of > 15 mm, or an extranodal lesion with a length diameter of > 10 mm according to PETCT or CT imaging;
5. For patients with B-ALL, the proportion of bone marrow primitive and naïve lymphocytes in the screening period ≥5%;
6. CD19 expression of tumor cells confirmed by flow cytometry or immunohistochemistry: the proportion of CD19 cells detected by peripheral blood flow cytometry in patients with B-ALL was ≥30%, and the proportion of CD19 cells in patients with B-cell lymphoma was positive by immunohistochemistry;
7. Adequate function of vital organs: liver function satisfies ALT≤3×ULN, AST≤3×ULN; serum creatinine≤140μmol/L; Total bilirubin ≤ 2× ULN, and total bilirubin ≤ 3.0× ULN for patients with Gilbert syndrome; Haemodynamically stable and left ventricular ejection fraction (LVEF) ≥45% as determined by echocardiography or multichannel radionuclide angiography (MUGA); No active pulmonary infection, transcutaneous arterial oxygen saturation ≥92% in non-oxygen-based state;
8. ECOG score: 0~2 points;
9. As judged by the investigator, the patient has an expected survival of more than 3 months;
10. Subjects of childbearing potential agree to use a reliable and effective method of contraception (excluding contraception during the safe period) for 2 years from the time of signing the informed consent form until receiving ECAR01 cell infusion.

Exclusion Criteria:

1. Episodes of central nervous system disease or presence of pathological changes within 6 months prior to screening, including but not limited to: stroke, stroke, aneurysm, epilepsy, convulsions, aphasia, severe head injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or mental disorder;
2. patients with B-ALL with confirmed diagnosis of isolated extramedullary recurrence;
3. presence of malignancies other than acute B-cell leukemia/B-cell lymphoma;
4. Received the following anti-tumor therapies before cell collection: chemotherapy, targeted therapy, and other drug therapy within 14 days or at least 5 half-lives; Radiotherapy within 14 days;
5. Vaccination, B-cell targeted therapy within 4 weeks prior to screening;
6. Patient has systemic autoimmune disease or immunodeficiency;
7. Grade 2~4 acute graft-versus-host disease (GVHD) or moderate to severe chronic GVHD within 4 weeks prior to screening;
8. Patients with relatively serious heart disease, such as angina, myocardial infarction, heart failure and arrhythmia;
9. History of severe allergy to drugs used in clinical studies or raw and excipient materials of experimental drugs, such as cyclophosphamide, fludarabine, DMSO, etc.;
10. Patient has active hepatitis B, or positive HCV antibody, or HIV antibody, or syphilis;
11. Presence of active infection requiring intravenous antibiotics or hospitalization;
12. Pregnant or lactating women;
13. Other investigators believe that the subject is not suitable to participate in this clinical study because it will affect the safety and efficacy judgment of the subject, or for other reasons;

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
1. Adverse events | up to 2 years
  Total number, incidence and severity of adverse events (AEs) in patients of ECAR01 infusion. The AEs will be assessed according to the 2019 Consensus on Cytokine Release Syndrome and Immune-cell-associated Neurotoxicity published by the American Society of Transplantation and Cell Therapy (ASTCT), the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 and EBMT 2019 consensus.

SECONDARY OUTCOMES:
2.The persistence, accumulation, and migration of CART cells | up to 2 years
  Assessing the trafficking of CART cells in the peripheral blood at the time of each infusion as well as at each time of follow-up by Quantitative Real-time Polymerase Chain Reaction or flow cytometry. Peripheral blood will be collected prior to the initial infusion and will be set as baseline.
Progression free survival (PFS) | up to 2 years
  Progression Free Survival (PFS) defined as the time from treatment to first documentation of objective leukemic progression (date of leukaemia assessment documenting progressive disease) or to death due to any cause. Progression is assessed by BM biopsy or CSF analysis according to NCCN criteria. It is assessed at Day 90 or earlier if clinically indicated.
Overall survival (OS) | up to 2 years
  Overall Survival (OS) defined as the time from treatment to the date of death due to any cause.
Objective Response Rate (ORR) | up to 2 years
  Overall response rate (ORR) is defined as proportion of participants who achieve overall response (CR/CRi).

CONTACTS AND LOCATIONS:
Overall Officials: bing xing wang, M.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, China

IPD SHARING:
Plan to Share IPD: Yes